CLINICAL TRIAL: NCT01829984
Title: A Comparison of Strategies for Injection Teaching: Verbal and Written Instruction Versus Verbal and Written Plus Simulation in Patients With Breast Cancer and Their Caregivers
Brief Title: Verbal and Written Instruction Versus Verbal and Written Plus Simulation in Patients With Breast Cancer and Their Caregivers
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 13-057
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Breast Cancer
Keywords: Injection Teaching; 13-057
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- control injection teaching: The first 25 subjects recruited into the study will be that control group. Subjects accrued during the control phase will receive the control injection teaching, which at MSKCC is verbal instruction. To minimize practice variation, the teaching will be provided by the office-practice nurse guided by a verbal script. The consented subjects will complete a questionnaire before the teaching, immediately after the teaching, and after performing the injection the following day. The nurse who administered the teaching will also complete an evaluation immediately following the teaching.
  Interventions: Other: Verbal and Written Instruction
- intervention group: The subsequent 25 subjects enrolled into the study will be in the intervention group. Subjects accrued during the intervention phase will receive the verbal and written injection teaching, plus demonstration and return demonstration using an injection model. It is anticipated that the intervention teaching will take no longer then 5 additional minutes, however time will be evaluated as a secondary objective as well in both groups. The consented subjects will complete a questionnaire before the teaching, immediately after the teaching, and after performing the injection the following day. The nurse who administered the teaching will also complete an evaluation immediately following the teaching.
  Interventions: Other: Verbal and Written Plus Simulation

INTERVENTIONS:
Other: Verbal and Written Instruction — Pre-teaching Evaluation: Patient
  * Pre-teaching Evaluation: Caregiver
    o To be completed immediately before the teaching. Administered by the nurse who will provide the teaching. The form utilized will depend on if the patient or caregiver will be administering the injection.
  * Post-teaching Evaluation: Patient Post-teaching Evaluation: Caregiver To be completed immediately after the teaching. Administered by the nurse who provided the teaching. The form utilized will depend on if the patient or caregiver will be administering the injection.
  Groups: control injection teaching
Other: Verbal and Written Plus Simulation — Post-injection Evaluation: Patient
  * Post-injection Evaluation: Caregiver
    o To be completed after the injection is administered (outside of MSKCC) by the patient or caregiver. The form utilized will depend on if the patient or caregiver has administered the injection. They will return this evaluation at the patient's next visit (2 weeks later).
  * Nurse Evaluation: Control
  * Nurse Evaluation: Model o To be completed immediately following the completion of the teaching by the nurse. The form utilized will depend on if the teaching was part of the control or intervention phase of the study.
  Groups: intervention group

SUMMARY:
The purpose of this study is to compare two different ways of teaching people how to give injections at home. The first is what we do now, which is teaching patients and/or their caregivers verbally and by giving written instructions. The second is what we do now (verbal and written instructions) along with a demonstration and practice using a needle and an injection pad that feels similar to skin and fat. This is being done to find the best method for teaching people to give an injection at home.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Over 18 years of age
* No history of performing injections
* Patient must be receiving pegfilgrastim during adjuvant or neoadjuvant chemotherapy
* Patient will have the pegfilgrastim administered at home either by self administering or by a caregiver.

Exclusion Criteria:

* Patient or caregiver desire to inject (with saline) during or immediately following the injection teaching
* Prior self-injection or injection administration experience of any type
* Patients with history of anaphylaxis or other severe reactions to latex
* Patients that required pegfilgrastim injection be administered in clinic

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All breast cancer medical oncology clinics at MSKCC will serve as recruitment clinics for the proposed study. Nurses will notify the PI of any patient due to start adjuvantadjuvant or neoadjuvant treatment when the regimen includes pegfilgrastim.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2013-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
compare verbal and written teaching for injection teaching | 1 year
  with verbal and written teaching + simulation using an injection model, in terms of:
  * Patient/caregiver satisfaction
  * Patient/caregiver self-confidence
  * Nurse satisfaction

SECONDARY OUTCOMES:
Assess for changes in patient self-reported | 1 year
  worry about injection before and after the injection teaching
Compare nurses' perceptions of patient/caregiver confidence levels | 1 year
  after injection teaching to actual patient/caregiver reported confidence levels
Compare the amount of nurses' time spent teaching | 1 year
  between the teaching modalities

CONTACTS AND LOCATIONS:
Overall Officials: Erica Fischer-Cartlidge, RN, MSN, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/